CLINICAL TRIAL: NCT03005808
Title: Choose Between Two Different Concentration of Ropivacaine on TAP Block for Children Submitted of Open Appendectomy
Brief Title: Choose the Best Concentration of Ropivacaine on TAP Block for Open Appendectomy in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Infantil Albert Sabin (Other)
Collaborators: Fortaleza University (Other)
Responsible Party: Principal Investigator, washington aspilicueta pinto filho, medical Anesthesiologist, Hospital Infantil Albert Sabin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HOSPITALIAS1
Record Dates: First submitted 2016-12-25; First posted 2016-12-29 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-12

CONDITIONS: Pain, Postoperative; Appendicitis
Keywords: appendectomy, pediatrics, nerve block, abdominal wall
MeSH Terms: conditions — Pain, Postoperative; Appendicitis | interventions — Ropivacaine; Appendectomy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control group (No Intervention): All patients had the same protocol of anesthesia and analgesia. The control group didn´t received block.
- TAP 0.25 group (Experimental): The TAP 0.25 group received TAP block with ropivacaine 0.25% 0.4ml/kg. All patients had the same protocol of anesthesia and analgesia.
  Interventions: Drug: Ropivacaine
- TAP 0.5 group (Experimental): The TAP 0.5 group received TAP block with ropivacaine 0.5% 0.4ml/kg. All patients had the same protocol of anesthesia and analgesia.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Surgery for appendicitis
  Other Names: Appendectomy
  Arms: TAP 0.25 group; TAP 0.5 group

SUMMARY:
Blockage of the transverse abdomen (TAP) promotes excellent analgesia of the abdominal wall and the parietal peritoneum. The TAP block could advange the postoperative pain of Appendectomy in children. The world literature doesn´t focus the best Ropivacaine´s concentration to improve postoperative pain in Appendectomy in children. We propose a randomized trial that compares 3 groups children submitted Appendectomy in children between 6 and 16 years. The control group has received no blockade, the other two groups have received TAP blocks if ropivacaine 0,25% and 0,5% 0.4ml/kg.

DETAILED DESCRIPTION:
Blockage of the transverse abdomen (TAP) promotes excellent analgesia of the abdominal wall and the parietal peritoneum. The meta-analyzes in adults demonstrate improved of postoperative pain and analgesic´s consumption. There are few studies on TAP block in open appendectomies and laparoscopic in pediatrics, they show good results. There is a consensus of the best anesthetic volume for good infiltration of the TAP block, but there are still doubts in the literature about the best concentration of local anesthetics of long duration. The main objective of this prospective, randomly distributed and double-blind clinical trial is to evaluate two concentrations of 0.25% and 0.5% ropivacaine with a volume of 0.4 ml / kg in pain control and the analgesic consumption through 24 hours observation in open Appendectomy in children between 6 and 16 years. 3 groups were being compared: the control group has received no blockade, the other two groups have received TAP blocks if ropivacaine 0,25% and 0,5% 0.4ml/kg. All pacients patients received the same protocols (anesthesia and analgesia). The provided analgesia was dipyrone every 6 hours and ketoprofen every 8 hours, and rescue analgesia was tramadol every 4hours if it were required. The FACE pain scale was used to evaluate the postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 and 16 years who were previously healthy submitted to appendectomy.

Exclusion Criteria:

* Children cardiac, pulmonary, renal and neurological diseases and allergy and refusal of parents, caregivers and patients to participate in the study.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2016-02 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Reduce the pain intensity using the Face Pain Scale | 24 hour after surgery
  Subjected to the same general anesthesia protocol and postoperative analgesia. The TAP0.25 and TAP0.5 groups received TAP block with ropivacaine 0.25% or 0.5% 0.4ml/kg, the control group didn´t receive block. The evaluation times were: 1 hour, 4 hours, 8 hours, 12 hours, 18 hours and 24 hours after surgery. The time elapsed was recorded, from the end of the surgery to the first use of tramadol. The parents and the patients themselves were instructed to request analgesic at any time.

SECONDARY OUTCOMES:
Reduce the opioid consumption through 24 hours postoperative observation | 24 hour after surgery
  Subjected to the same general anesthesia protocol and analgesia. The TAP0.25 and TAP0.5 groups received TAP block with ropivacaine 0.25% or 0.5% 0.4ml/kg, the control group didn´t receive block. All patients received dipyrone and ketoprofen, the rescue analgesic used was tramadol 1.5mg / kg (maximum dose of 100mg) up to 4 / 4h when Face´s Scales reached 5 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Infantil Albert Sabin, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abu Elyazed MM, Mostafa SF, Abdullah MA, Eid GM. The effect of ultrasound-guided transversus abdominis plane (TAP) block on postoperative analgesia and neuroendocrine stress response in pediatric patients undergoing elective open inguinal hernia repair. Paediatr Anaesth. 2016 Dec;26(12):1165-1171. doi: 10.1111/pan.12999. Epub 2016 Oct 12. PMID 27731956
- [Background] Carney J, Finnerty O, Rauf J, Curley G, McDonnell JG, Laffey JG. Ipsilateral transversus abdominis plane block provides effective analgesia after appendectomy in children: a randomized controlled trial. Anesth Analg. 2010 Oct;111(4):998-1003. doi: 10.1213/ANE.0b013e3181ee7bba. Epub 2010 Aug 27. PMID 20802056
- [Background] Lapmahapaisan S, Tantemsapya N, Aroonpruksakul N, Maisat W, Suraseranivongse S. Efficacy of surgical transversus abdominis plane block for postoperative pain relief following abdominal surgery in pediatric patients. Paediatr Anaesth. 2015 Jun;25(6):614-20. doi: 10.1111/pan.12607. Epub 2015 Jan 9. PMID 25571981
- [Background] Reinoso-Barbero F, Poblacion G, Builes LM, Castro LE, Lahoz AI. Successful ultrasound guidance for transversus abdominis plane blocks improves postoperative analgesia after open appendicectomy in children. Eur J Anaesthesiol. 2012 Aug;29(8):402-4. doi: 10.1097/EJA.0b013e328353570e. No abstract available. PMID 22488336